CLINICAL TRIAL: NCT01784822
Title: Zenapro™ Hybrid Hernia Repair Device for Ventral Hernia Repair
Status: Completed | Type: Observational
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-013
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Ventral Hernias
Keywords: Ventral hernia; Graft repair
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (1):
- Zenapro™ Hybrid Hernia Repair Device: Device to be used to reinforce or bridge the abdominal wall for the repair of ventral hernias.
  Interventions: Device: Zenapro™ Hybrid Hernia Repair Device

INTERVENTIONS:
Device: Zenapro™ Hybrid Hernia Repair Device — Device will be placed during open or laparoscopic hernia repair.

SUMMARY:
The objective this study is to collect post-market data on the performance of the Zenapro™ Hybrid Hernia Repair Device when used to reinforce or bridge the abdominal wall for the repair of ventral hernias.

ELIGIBILITY:
Inclusion Criteria:

* Primary or recurrent ventral hernia
* Need for abdominal wall repair with reinforcement or bridging material to obtain the desired surgical result

Exclusion Criteria:

* Age < 21 (i.e., infants, children)
* Device intended to be used in an infected wound
* Known sensitivity to porcine material
* Pregnant or planning pregnancy in the future
* Life expectancy of less than 12 months from the date of the index procedure
* Hernia too large to be covered with a single device with at least 4-5 cm of tissue overlap on all sides

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from University of Tennessee, Duke University and Cleveland Clinic
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2013-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Rate of hernia recurrence | 12 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Tennessee, Knoxville, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia